CLINICAL TRIAL: NCT04969146
Title: A Sleep Intervention for Cancer Patients and Their Caregivers
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jennifer Steel, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY19090202
Record Dates: First submitted 2021-07-16; First posted 2021-07-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intervention; Control
Keywords: Sleep Quality; Depression; Quality of Life; Dyadic Function
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups receiving different interventions in parallel for the duration of the study
Who Masked: Investigator
Masking Description: Research Coordinators will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Cognitive Behavioral Therapy Intervention Dyadic (Experimental): The patient and caregiver in the dyadic intervention will have 5 sessions of Modified CBTi. The patient and caregiver will complete the assessment at 3- and 6 months follow up.
  Interventions: Behavioral: Dyadic Intervention
- Modified Cognitive Behavioral Therapy Intervention Patient Only (Experimental): The patient in the patient only intervention arm will receive 5 sessions of Modified CBTi. The patient and caregiver will complete the assessment at 3- and 6 months follow up
  Interventions: Behavioral: Patient Only Intervention

INTERVENTIONS:
Behavioral: Dyadic Intervention — The patient and caregiver dyads will complete and return baseline questionnaires and then be randomized to Modified CBTi Dyadic Intervention. The patient and caregiver in the dyadic intervention will have 5 sessions of Modified CBTi. Upon completion of the intervention, the patient and caregiver will complete the follow up assessments at approximately 3 months and 6 months after the baseline questionnaires.
  Arms: Modified Cognitive Behavioral Therapy Intervention Dyadic
Behavioral: Patient Only Intervention — The patient and caregiver dyads will complete and return baseline questionnaires and then be randomized to Modified CBTi Patient Only Intervention. The patient in the Patient Only Intervention will have 5 sessions of Modified CBTi. Upon completion of the intervention, the patient and caregiver will complete the follow up assessments at approximately 3 months and 6 months after the baseline questionnaires.
  Arms: Modified Cognitive Behavioral Therapy Intervention Patient Only

SUMMARY:
The purpose of the study is to design and test a dyadic sleep intervention for patients diagnosed with cancer and their intimate partner.

DETAILED DESCRIPTION:
Sleep problems remain underdiagnosed and undertreated among cancer patients despite their high prevalence and consequences to quality of life and health. Hepatobiliary cancer patients have one of the highest rates of sleep problems with 59% reporting poor sleep quality and 43% reporting sleeping less than 6 hours per night. Sleep problems were found to be associated with clinical levels of depressive symptoms, elevations in pain and fatigue. Investigators have observed that short sleep duration was associated with increased risk of mortality in patients with hepatobiliary cancers. Inflammation has been hypothesized to mediate the link between sleep and mortality. In hepatobiliary cancer, short sleep duration was associated with elevations in Interleukin (IL)-6, IL-1, IL-1 and IL-2 and poor sleep quality with elevations in Interferon (IFN) Interleukin-2, after adjusting for tumor associated inflammation, mediated the link between sleep duration and survival. These pro-inflammatory cytokines are also related to tumor growth and development of metastases. Sleep problems of spouses or intimate partners of hepatobiliary cancer patients were also prevalent with 62% reporting poor sleep quality and 33% reporting sleep less than 6 hours per night. Caregiving for an intimate partner with cancer has been linked to increased mortality and sleep has been proposed as a possible mediator of this link. Face to face cognitive behavioral therapy (CBT) has been shown to be effective in cancer patients and cancer caregivers. However, due to the distance patients travel to our medical center (58% >1 hour), infrequency of visits (e.g., approximately every two months), limited resources (48% of patients <$20,000 annual income), and the unpredictability of cancer-related symptoms; weekly face-to- face CBT to treat sleep problems is not feasible. Therefore, investigators will test a dyadic Modified Cognitive Behavioral Therapy for Insomnia (CBTi) intervention to reduce insomnia in patients and possibly caregivers and expect the findings of this study to have a significant public health impact for the over 12 million cancer patients and spousal/partner caregivers in which nearly half are estimated to suffer from sleep problems.

ELIGIBILITY:
Inclusion Criteria:

Patient

* Diagnosed with cancer
* Screens positive for sleep problems (5 or greater score on the PSQI)
* Shares a bed with the caregiver/intimate partner
* Patient's caregiver/intimate partner also screens positive for sleep problems (5 or greater score on the PSQI)

Exclusion Criteria:

Patient or Caregiver

* does not screen positive for sleep problems
* has been diagnosed with sleep apnea or use a continuous positive airway pressure (CPAP) machine
* has been diagnosed with narcolepsy or restless legs
* works in a job that requires shift changes
* does not speak/read English
* does not share a bed with intimate partner

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2027-08-16 (Estimated); Primary Completion 2028-12-23 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Change from baseline in insomnia reduction at 6 months
  Insomnia Reduction by 50% -Total Score (0-28, where 28 is most severe)
Insomnia Severity Index | Change from baseline in insomnia reduction at 12 months
  Insomnia Reduction by 50% -Total Score (0-28, where 28 is most severe)

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline in improved sleep latency at 6 months.
  Improved Sleep Latency by 25% - Global Score ranging from 0 to 21, where lower score indicates better quality of sleep
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline in improved sleep latency at 12 months
  Improved Sleep Latency by 25% - Global Score ranging from 0 to 21, where lower score indicates better quality of sleep
Patient-reported Outcomes Measurement Information System (PROMIS-29) | Change from baseline in improved quality of life at 6 months
  Increase in Quality of Life by 25% - total score ranging from 20-80, where lower scores indicate better quality of life
Patient-reported Outcomes Measurement Information System (PROMIS-29) | Change from baseline in improved quality of life at 12 months
  Increase in Quality of Life by 25% - total score ranging from 20-80, where lower scores indicate better quality of life

OTHER OUTCOMES:
Patient-reported Outcomes Measurement Information System (PROMIS-29) | Change from baseline in depressive symptoms at 6 months
  Reduction of Depressive Symptoms by 25%- total score ranging from 20-80, where lower scores indicate better quality of life
Patient-reported Outcomes Measurement Information System (PROMIS-29) | Change from baseline in depressive symptoms at 12 months
  Reduction of Depressive Symptoms by 25%- total score ranging from 20-80, where lower scores indicate better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Steel, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center Montefiore Liver Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified Data may be shared with investigators who request data from the Primary Investigator
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the end of the study for up to one year.
Access Criteria: Appropriate investigator credentials (MD, PhD) and request, and for up to one year after study completion